CLINICAL TRIAL: NCT05461963
Title: Breastfeeding and Miscarriage Relationship
Brief Title: The Relationship Between Breastfeeding During Early Pregnancy and Miscarriage
Status: Completed | Type: Observational
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Serif Aksin, associate professor, Siirt University
Other Study IDs: SiirtUN
Record Dates: First submitted 2022-06-26; First posted 2022-07-18 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Miscarriage; Breast Feeding
MeSH Terms: conditions — Abortion, Spontaneous; Breast Feeding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- breastfeeding pregnants( n:76): pregnants in early weeks of pregnancy who practice breastfeeding
- control group ( n:76): pregnants in early weeks of pregnancy who not practice breastfeeding

SUMMARY:
Breastfeeding provides various health and psychological benefits to mothers and their babies. It also acts as an effective method of natural contraception when applied strictly for up to six months after birth. Studies show that breastfeeding times are getting longer in the USA and more babies are breastfed for more than 12 months compared to the past. Recent research shows that 57% of US infants are breastfed until at least six months of age, and more than a third continue to be breastfed for up to 12 months. Prolonged breastfeeding durations increase the prevalence of breastfeeding during pregnancy, especially with the shortening of the intervals between pregnancies. Breastfeeding during pregnancy is a relatively common practice in many parts of the world. According to the data of studies conducted in low- and middle-income countries, it has been determined that 35% of the last born babies continue to be breastfed in the next pregnancy of their mothers. It has also been shown that the prevalence of breastfeeding during pregnancy in low-income countries is between 15% and 50%. Few research has been done on the relationship between breastfeeding during pregnancy and maternal, infant, or pregnancy outcomes. Some studies have suggested that hormonal mechanisms in pregnancy may link breastfeeding during pregnancy and abortion. When babies stimulate the nipple and areola during sucking, they trigger the release of oxytocin in the mother, causing a series of reactions that push the milk towards the nipple. We know that the prevalence of short and long breastfeeding intervals in pregnancy is high in our country. Therefore, in this study, we are planning to investigate whether there is a relationship between breastfeeding during pregnancy and miscarriage based on this information.

DETAILED DESCRIPTION:
Our aim in this study is to investigate whether breastfeeding during pregnancy increases the risk of abortion and to determine whether there is a relationship between them. For this purpose, approximately 76 pregnant women who were pregnant and continuing to breastfeed in Siirt Training and Research Hospital between June 2022 and December 2022 will be included in the study. The same number (n:76) non-breastfeeding pregnant control group will be included in the study. Age, gestational week, pregnancy history (gravida, parity, abortion, missed, ectopic),breastfeeding time in previous pregnancies, bleeding, daily breastfeeding frequency and medical history of the pregnant will be recorded. In the light of the information obtained in this way, we plan to determine whether there is a relationship between breastfeeding during pregnancy and abortion.

ELIGIBILITY:
Inclusion Criteria:

* being breastfeeding
* being at the 1.st trimester of pregnancy

Exclusion Criteria:

* history of inherited thrombophilia
* history of uterine anomaly
* history of trauma
* history of genetic anomaly
* history of habitual abortus

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant women over the age of 18 who are in the first trimester of pregnancy and continue to breastfeed
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Miscarriage, ratio in breastfeeding pregnant women | From the 6th week of pregnancy to the 20th week.
  Miscarriage is the spontaneous loss of a pregnancy before the 20th week,

CONTACTS AND LOCATIONS:
Overall Officials: Şerif Aksin, Study Director — Siirt University Medical Faculty Obstetrics and Gynecology Departmant
Locations (1):
- Siirt Üniversity Medical Faculty, Siirt, Turkey (Türkiye)

REFERENCES:
- [Background] Molitoris J. Breast-feeding During Pregnancy and the Risk of Miscarriage. Perspect Sex Reprod Health. 2019 Sep;51(3):153-163. doi: 10.1363/psrh.12120. Epub 2019 Sep 16. PMID 31524957
- [Background] Lopez-Fernandez G, Barrios M, Goberna-Tricas J, Gomez-Benito J. Breastfeeding during pregnancy: A systematic review. Women Birth. 2017 Dec;30(6):e292-e300. doi: 10.1016/j.wombi.2017.05.008. Epub 2017 Jun 19. PMID 28642112
- [Background] Ayrim A, Gunduz S, Akcal B, Kafali H. Breastfeeding throughout pregnancy in Turkish women. Breastfeed Med. 2014 Apr;9(3):157-60. doi: 10.1089/bfm.2013.0086. Epub 2013 Oct 25. PMID 24160359